CLINICAL TRIAL: NCT04531735
Title: Is Respiratory Syncytial Virus Infection More Dangerous Than Covid 19 in the Neonatal Period?
Brief Title: Respiratory Syncytial Virus Infection May be More Dangerous in Neonate
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Dr. Behcet Uz Children's Hospital (Other)
Responsible Party: Principal Investigator, Senem Alkan Özdemir, Associate Professor of Neonatology, Dr. Behcet Uz Children's Hospital
Other Study IDs: 2020/522
Record Dates: First submitted 2020-08-19; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: RSV Infection; Covid19
Keywords: newborn; covid infection; viral infection; RSV infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; COVID-19; Virus Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: COVID positive infants
- Group 2: RSV positive infants

SUMMARY:
Investigators aimed to compare clinical and radiographic markers between SARS-CoV-2 positive and RSV positive infants

DETAILED DESCRIPTION:
This single center cross-sectional study was conducted in University of Health Sciences Dr Behçet Uz Children's Hospital with a 400-bed tertiary care hospital in İzmir, Turkey, during the period of March 11 - April 30, 2020. This hospital is a pediatric referral center in the Aegean Region of Turkey with annual approximately 600,000 outpatients and 24,000 hospitalizations. All children with fever and cough who were tested by taken nasopharyngeal swabs for SARS-CoV2 and common human respiratory tract pathogens were included in the study.

The clinician responsible for taking the respiratory samples were trained by the infection control committee on sampling and using personal protective equipment. Firstly, an oropharyngeal sampling was taken, and then a nasopharyngeal sampling was taken using the same swab from patient with fever and cough/shortness of breath for SARS-CoV-2 PCR. The same swab was used and placed in the same transport medium. The samples were sent to the laboratory determined by the Ministry of Health, following the cold chain rules. The protocol of Real Time-PCR was consistent with the recommendation of the WHO. Real time-PCR was performed at the local governmental centers for disease control and prevention. The kit wasapplied to nucleic acid isolates from nasopharyngeal aspirate/lavage, bronchoalveolar lavage, nasopharyngeal swab, oropharyngeal swab and sputum samples. Rapid diagnosis with the kit is achieved via one-step reverse transcription (RT) and real-time PCR (qPCR) (RT-qPCR) targeting SARS-CoV-2 (2019-nCoV)-specific RNA-dependent RNA polymerase (RdRp) gene fragment. The RdRp gene-targeted Wuhan-RdRp oligonucleotide set gives positive results only with SARS-CoV-2 (2019-nCoV)( Bio-Speedy®, Turkey SARS-CoV-2 (2019-nCoV) qPCR Detection Kit)

Respiratory samples taken by nasopharyngeal swabs were tested for common human respiratory tract pathogens. For the testing of samples, real-time polymerase chain reaction (PCR) assay was performed. In the assay a commercial multiplex real-time PCR kit (Bosphore Respiratory Pathogens Panel Kit V4, Anatolia Geneworks, Turkey) was used to investigate the presence of Influenza viruses ( Influenza A, Pandemic H1N1 Influenza A, Seasonal H1N1 Influenza A and Influenza B), Parainfluenza (PIV) viruses (PIV-1, PIV-2, PIV-3 and PIV-4), Human Coronaviruses (HCoV) (CoV OC43, CoV NL63, CoV HKU1 and CoV 229E), Respiratory Syncytial Virus (RSV) A/B, Rhinovirus, Metapneumovirus, Enterovirus, Bocavirus, Adenovirus, Parechovirus and bacterial pathogens such as Mycoplasma pneumonia, Moraxella catarrhalis, Bordetella pertussis and Haemophilus influenzae type B in the clinical samples.

Demographic, epidemiological and clinical data were obtained from hospital electronic information system medical records. For the statistical evaluation of the data, SPSS 20.0 Microsoft for Windows (IBM Corporation, Armonk, NY, USA). was used and P <0.05 value was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

During the study period respiratory symptoms at the NICU admission will be included

Exclusion Criteria:

Congenital abnormalities

Ages: 4 Days to 1 Month | Sex: All
Age Groups: Child
Study Population: Newborns with respiratory symptoms
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Oxygen status and evaluation of neonatal intensive care stay | 3 months
  Total neonatal intensive care duration, total duration of oxygen supplement

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Behçet Uz Children's Hospital, İzmirli, İzmir
  - İzmir Dr. Behcet Uz Training and Research Hospital, Izmir

IPD SHARING:
Plan to Share IPD: No